CLINICAL TRIAL: NCT06684678
Title: Efficacy of Individualized Automatic Coaching Message Based on the Metrics of Continuous Glucose Monitoring and Depressive Symptom: A Randomized Controlled Trial
Brief Title: Individualized Automatic Coaching Message for Glycemic Management and Depressive Symptom
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Gyuri Kim, Principal Investigator, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SamsungMC_ENDO_2; SMO124027 (Other Grant/Funding Number: Samsung Medical Center); 2024F-2 (Other Grant/Funding Number: Korean Diabetes Association); RS-2024-00399025 (Other Grant/Funding Number: Korea Health Industry Development Institute (KHIDI))
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 1; Continuous Glucose Measurement
Keywords: type 1 diabetes; continuous glucose monitoring; depressive symptom
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Depression

STUDY DESIGN:
Intervention Model Description: 1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized automatic coaching message for glycemic management and depressive symptoms (Experimental): The study will enroll patients with type 1 diabetes who are already receiving twice-monthly non-face-to-face management by a dedicated education nurse through the Type 1 Diabetes Home Care Project and Educational Consultation program. For 12 weeks, the intervention group will receive weekly personalized coaching messages for glycemic management based on data from continuous glucose monitoring and bi-weekly personalized coaching messages for depression symptoms based on depression questionnaires, instead of non-face-to-face diabetes management.
  Interventions: Other: individualized automatic coaching message for glycemic management and depressive symptom
- Current Treatment (No Intervention): The study will enroll patients with type 1 diabetes who are already receiving twice-monthly non-face-to-face management by a dedicated education nurse through the Type 1 Diabetes Home Care Project and Educational Consultation program. The control group will continue their current treatment and non-face-to-face diabetes management.

INTERVENTIONS:
Other: individualized automatic coaching message for glycemic management and depressive symptom — For 12 weeks, the intervention group will receive weekly personalized coaching messages for glycemic management based on data from continuous glucose monitoring and bi-weekly personalized coaching messages for depression symptoms based on depression questionnaires, instead of non-face-to-face diabetes management.
  Arms: Individualized automatic coaching message for glycemic management and depressive symptoms

SUMMARY:
This is a single-center, randomized, prospective, confirmatory study of efficacy of individualized automatic coaching message for glycemic management and depressive symptom in patients with type 1 diabetes. The study will enroll patients with type 1 diabetes who are applying continuous glucose monitoring (CGM) and receiving twice-monthly non-face-to-face management by a dedicated education nurse through the Type 1 Diabetes Home Care Project and Educational Consultation program. For 12 weeks, the intervention group will receive weekly personalized coaching messages for glycemic management based on data from continuous glucose monitoring and bi-weekly personalized coaching messages for depression symptoms based on depression questionnaires, instead of non-face-to-face diabetes management. The control group will continue their current treatment and non-face-to-face diabetes management. The aim of this study is to evaluate whether the efficacy of automated, personalized coaching messages for glycemic management and depressive symptoms is non-inferior to the current non-face-to-face management approach in people with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes, age 18-75 years old
* Patients who have used continuous glucose monitoring at least three months and have enrolled in Type 1 Diabetes Home Care Project and Educational Consultation program.
* Patients with at least 70% of 14 days of continuous glucose monitor data within the past month
* Glycated hemoglobin 7% or higher, or Glycated hemoglobin 6% or higher but less than 7% and failing to meet 1 of the continuous glucose monitor blood glucose target values: time in range (70-180 mg/L) 70% or less, or time below range (<70 mg/L) 4% or more, or time above range (>180 mg/L) 25% or more, or glucose management indicator (GMI) 7% or more, or coefficient of variation (CV%) 36% or more.
* Currently receiving treatment with multiple insulin injection therapy
* Patients who have access to KakaoTalk via smartphone and are able to communicate with it
* Voluntarily agreed to participate in this clinical study.

Exclusion Criteria:

* Steroid and immunosuppressant users. But it can be included if patients continuously maintain same drug dose at least three months.
* Breastfeeding or pregnant patients
* Patients who do not voluntarily consent to the study
* Anyone deemed unsuitable by the investigator to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-11-13 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Time In Range | Week 12
  Derived from continuous glucose monitoring (CGM)

SECONDARY OUTCOMES:
Diabetes treatment satisfaction | Week 12
  Diabetes Treatment Satisfaction Questionnaire (DTSQ);
  Minimum and Maximum Values: The DTSQ consists of eight items, with six items measuring satisfaction scored on a 0-6 scale (where 0 is very dissatisfied and 6 is very satisfied). The scores for these six items are summed, giving a total score range from 0 to 36.
  Higher Scores: Higher scores on the DTSQ indicate better satisfaction with diabetes treatment. A higher total score suggests greater satisfaction, while a lower score indicates dissatisfaction.
Depressive symptoms | Week 12
  Patient Health Questionnaire-9 (PHQ-9); Minimum and Maximum Values: The PHQ-9 consists of nine items, each scored from 0 (not at all) to 3 (nearly every day). The scores for each item are summed to give a total score, resulting in a range from 0 to 27.
  Higher Scores: Higher scores on the PHQ-9 indicate worse outcomes, meaning greater severity of depressive symptoms. Lower scores suggest fewer symptoms of depression or none at all.
  Interpretation of Scores:
  0-4: Minimal or no depression; 5-9: Mild depression; 10-14: Moderate depression; 15-19: Moderately severe depression; 20-27: Severe depression
Time In Tight Range | Week 12
  Derived from CGM
Level of Glycated Hemoglobin | Week 12
  Derived from blood measurement
Time Above Range | Week 12
  Derived from CGM
Time Below Range | Week 12
  Derived from CGM
Coefficient of Variation | Week 12
  Derived from CGM
Glycemic Management Indicator | Week 12
  Derived from CGM

OTHER OUTCOMES:
Level of Albuminuria | Week 12
  Urine creatinine-to-albumin ratio
Level of Glycated albumin | Week 12
  Glycated albumin
Level of total cholesterol | Week 12
  total cholesterol from blood measurement
Level of triglycerides | Week 12
  Level of triglycerides from blood measurement
Level of HDL (high density lipoprotein) cholesterol | Week 12
  Level of HDL cholesterol from blood measurement
Level of LDL (low density lipoprotein) cholesterol | Week 12
  Level of LDL cholesterol from blood measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No